CLINICAL TRIAL: NCT06309914
Title: The Effects of Indena's Mirtoselect® Bilberry Extract, Virtiva® Ginkgo Biloba Extract, and Enovita® Grape Seed Extract on Cognitive Performance and Mood States Over a 4-week Time Course
Brief Title: The Effects of Mirtoselect®, Virtiva®, and Enovita® on Cognitive Performance and Mood States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00074459
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Mental Processes; Cognitive Change; Mood Change
Keywords: Bilberry Extract; Ginkgo Biloba Extract; Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): One dose (1 capsule) will be consumed twice daily for 28 days. The placebo product will be rice flour (other ingredients: hypromellose, magnesium stearate and chlorophyll). Its appearance will be green/green oblong veggie capsule with white to off-white powder fill.
  Interventions: Dietary Supplement: Placebo
- Enovita Dietary Supplement (Experimental): One dose (1 capsule) will be consumed twice daily for 28 days. A single dose contains: 150mg grape seed extract (Vitis vinifera L) and dried seed (cultivated), and 27.50mg 95% polyphenols.
  Interventions: Dietary Supplement: Enovita Grape Seed Extract
- Mirtoselect Dietary Supplement (Experimental): One dose (1 capsule) will be consumed twice daily for 28 days. A single dose contains: 160mg bilberry extract (Vaccinium myrtillus L.) and 57.6mg 36% anthocyanosides.
  Interventions: Dietary Supplement: Mirtoselect Bilberry Extract
- Virtiva Dietary Supplement (Experimental): One dose (1 capsule) will be consumed twice daily for 28 days. A single dose contains: 240mg Ginkgo biloba extract (leaf), 28.8mg 12% phosphatidylserine (from sunflower), and 12mg 5% ginkgo flavonglycosides.
  Interventions: Dietary Supplement: Virtiva Plus Ginko Biloba Extract

INTERVENTIONS:
Dietary Supplement: Placebo — Subjects will consume one capsule of the Placebo twice daily for 28 days. At Day 0, they will perform the full cognitive assessment (~45 minutes) and complete the abbreviated POMS questionnaire in a fasted state. Immediately after, subjects will consume two capsules of their randomly assigned study product. At 60 minutes post-consumption, subjects will repeat the computerized cognitive assessment. At 180 minutes post-consumption, subjects will repeat the computerized cognitive assessment and abbreviated POMS questionnaire. Subjects will then be instructed to continue to take their respective study product twice daily, one capsule with the first meal of the day and one capsule with the evening meal, for the duration of the supplementation period (28 days). After 28 days of supplementation, subjects will be reassessed on the computerized cognitive assessment and abbreviated POMS.
  Arms: Placebo
Dietary Supplement: Enovita Grape Seed Extract — Subjects will consume one capsule of Enovita twice daily for 28 days. At Day 0, they will perform the full cognitive assessment (~45 minutes) and complete the abbreviated POMS questionnaire in a fasted state. Immediately after, subjects will consume two capsules of their randomly assigned study product. At 60 minutes post-consumption, subjects will repeat the computerized cognitive assessment. At 180 minutes post-consumption, subjects will repeat the computerized cognitive assessment and abbreviated POMS questionnaire. Subjects will then be instructed to continue to take their respective study product twice daily, one capsule with the first meal of the day and one capsule with the evening meal, for the duration of the supplementation period (28 days). After 28 days of supplementation, subjects will be reassessed on the computerized cognitive assessment and abbreviated POMS.
  Arms: Enovita Dietary Supplement
Dietary Supplement: Mirtoselect Bilberry Extract — Subjects will consume one capsule of Mirtoselect twice daily for 28 days. At Day 0, they will perform the full cognitive assessment (~45 minutes) and complete the abbreviated POMS questionnaire in a fasted state. Immediately after, subjects will consume two capsules of their randomly assigned study product. At 60 minutes post-consumption, subjects will repeat the computerized cognitive assessment. At 180 minutes post-consumption, subjects will repeat the computerized cognitive assessment and abbreviated POMS questionnaire. Subjects will then be instructed to continue to take their respective study product twice daily, one capsule with the first meal of the day and one capsule with the evening meal, for the duration of the supplementation period (28 days). After 28 days of supplementation, subjects will be reassessed on the computerized cognitive assessment and abbreviated POMS.
  Arms: Mirtoselect Dietary Supplement
Dietary Supplement: Virtiva Plus Ginko Biloba Extract — Subjects will consume one capsule of Virtiva Plus twice daily for 28 days. At Day 0, they will perform the full cognitive assessment (~45 minutes) and complete the abbreviated POMS questionnaire in a fasted state. Immediately after, subjects will consume two capsules of their randomly assigned study product. At 60 minutes post-consumption, subjects will repeat the computerized cognitive assessment. At 180 minutes post-consumption, subjects will repeat the computerized cognitive assessment and abbreviated POMS questionnaire. Subjects will then be instructed to continue to take their respective study product twice daily, one capsule with the first meal of the day and one capsule with the evening meal, for the duration of the supplementation period (28 days). After 28 days of supplementation, subjects will be reassessed on the computerized cognitive assessment and abbreviated POMS.
  Arms: Virtiva Dietary Supplement

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 4-week intervention clinical study assessing the efficacy of Mirtoselect®, Virtiva® Plus, and Enovita® on cognitive performance and mood states, and the occurrence of adverse events in response to daily supplementation. The desired sample size for this study is 64 subjects. To account for potential dropouts, we aim to enroll up to 20% over the desired sample size. Therefore, this study will enroll up to 76 healthy men and women (25-55 years of age). Subjects will be randomly divided into four study groups: Placebo, Virtiva® ginkgo biloba extract, Mirtoselect® bilberry extract, or Enovita® grape seed extract. Blocked randomization will be deployed in which subjects are divided into blocks of 4 subjects and each subject within a block is randomly assigned to one of the four study groups.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 4-week intervention clinical study assessing the efficacy of Mirtoselect®, Virtiva® Plus, and Enovita® on cognitive performance and mood states, and the occurrence of adverse events in response to daily supplementation. The desired sample size for this study is 64 subjects. To account for potential dropouts, we aim to enroll up to 20% over the desired sample size. Therefore, this study will enroll up to 76 healthy men and women (25-55 years of age). Subjects will be randomly divided into four study groups: Placebo, Virtiva® ginkgo biloba extract, Mirtoselect® bilberry extract, or Enovita® grape seed extract. Blocked randomization will be deployed in which subjects are divided into blocks of 4 subjects and each subject within a block is randomly assigned to one of the four study groups. There are 4 study events for this trial as follow:

Event 1 - Pre-screening/enrollment (Day -30 to Day -1): The potential subject will present a health history questionnaire to screen for study eligibility described in sections 5.2.1 (inclusion criteria) and 5.2.2 (exclusion criteria). The questionnaire will be reviewed by the Investigator or designee, and if the subject is eligible, they will be presented with an IRB approved ICF. The potential subject will be given the opportunity to review the ICF, ask any questions they may have to the Investigator or designee, and will be allowed to take the ICF home for review. The potential subject will be required to sign the ICF for study enrollment to proceed with study participation.

Event 2 - Familiarization with study procedures (computerized cognitive testing, questionnaires, and adverse event report) (Day -7 to Day -1): After obtaining written informed consent form the subject they will be scheduled for familiarization. At familiarization subjects will provide demographic details and will be assessed for anthropometrics (height, weight, body mass index). Subjects will undergo an abbreviated version (~15 minutes) of the computerized cognitive testing to familiarize with the online platform, testing instructions, and cadence of the tests. Subjects will be shown a clean copy of the abbreviated Profile of Mood States (POMS) questionnaire and the Investigator or designee will describe the questionnaire and provide instructions for completing the questionnaire. The Investigator or designee will explain adverse event reporting and instruct the subject to notify the research staff immediately, or as soon as possible, after the onset of any adverse event. After completion of the familiarization procedures, subjects will be randomly assigned to one of four study groups (Placebo, Virtiva® ginkgo biloba extract, Mirtoselect® bilberry extract, or Enovita® grape seed extract) and will be assigned a subject No./ID in the 100 series starting with "101" and continuing in sequential order until enrollment is met.

Event 3 - Baseline assessment (Day 0): In a fasted state, subjects will perform the full computerized cognitive assessment (~45 minutes) and complete the abbreviated POMS questionnaire (Pre). Immediately after, subjects will consume two capsules of their randomly assigned study product. At 60-minutes post consumption, subjects will repeat the computerized cognitive assessment and will be queried for adverse events. At 180-minutes post consumption, subjects will repeat the computerized cognitive assessment followed by the abbreviated POMS questionnaire, and will be queried for adverse events. The intent of the 60- and 180-minute follow up testing is to investigate potential acute effects of the study products. After the completion of Day 0, subjects will be instructed to continue to take their respective study product twice daily, one capsule with the first meal of the day and one capsule with the evening meal, for the duration of the supplementation period (28 days).

Event 4 - Final Post-Testing (Day 29 to Day 31): After 28 days of supplementation, subjects will be reassessed on the computerized cognitive assessment, abbreviated POMS, and queried for adverse events. Following these assessments, the subjects will have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 to 55 years
* Willing and able to give written informed consent
* Able to read, understand, sign and date the informed consent document (English only)
* Able and willing to comply with the schedule visit(s) and study requirements.

Exclusion Criteria:

* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirements and/or record the necessary study measurements.
* History of cardiovascular disease
* History of neurological disorders
* History of gastrointestinal disorders that could lead to uncertain absorption of the study supplements
* History of kidney or liver disease
* History of metabolic disorders (diabetes, metabolic syndrome, other)
* History or current malignancy
* Receiving chemotherapy agents or radiation treatments
* Diagnosis of a terminal illness
* Pregnancy or has breastfed within 3 months prior to enrollment
* Use of prescription medications that impact digestion
* History or current alcohol or drug abuse
* Has significant concurrent illnesses (controlled or uncontrolled)
* Participation in any other investigational study within 30 days prior to consent

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Change in Visual Memory | Baseline, Day 28
  The visual memory test measures how well a subject can recognize, remember, and retrieve geometric figures or spatial representations.
Change in Verbal Memory | Baseline, Day 28
  The verbal memory test measures how well a subject can recognize, remember, and retrieve words.
Change in Finger Tapping Test (FTT) Results | Baseline, 60 mins post-supplementation on day 0, 180 mins post-supplementation on Day 0, and Day 28.
  The FTT measures the speed and number of finger-taps on each hand. This tests the motor speed and fine motor capability of subjects.
Change in Symbol Digit Coding (SDC) Test Results | Baseline, 60 mins post-supplementation on day 0, 180 mins post-supplementation on Day 0, and Day 28.
  Measures the speed of processing while drawing upon several cognitive processes simultaneously (i.e., visual scanning, visual perception, visual memory, and motor functions).
Change in Stroop Test Results | Baseline, 60 mins post-supplementation on day 0, 180 mins post-supplementation on Day 0, and Day 28.
  Assesses the ability to inhibit cognitive interference that occurs when the processing of a stimulus impedes the simultaneous processing of a second stimulus.
Change in Shifting Attention Test Results | Baseline, 60 mins post-supplementation on day 0, 180 mins post-supplementation on Day 0, and Day 28.
  Measures a subject's executive function (i.e., rules, categories, decision making) or their ability to shift from one instruction set to another quickly and accurately.
Change in Continuous Performance Test Results | Baseline, 60 mins post-supplementation on day 0, 180 mins post-supplementation on Day 0, and Day 28.
  Measures vigilance or sustained attention over time.

SECONDARY OUTCOMES:
Change in Abbreviated Profile of Mood States (POMS) Score | Baseline, 60 mins post-supplementation on day 0, 180 mins post-supplementation on day 0, and Day 28.
  Changes assessed in the abbreviated profile of mood states for subjective assessment of the subject's mood and overall well-being. It is a 40 point scale, divided into 7 different subscales, with a 5 point Likert scale, ranging from 0 (not at all) to 4 (Extremely) of how a subject feels in response to that particular feeling. The following equation is used to determine the overall score: Total Mood Disturbance = [Tension+Depression+Anger+Fatigue+Confusion] - [Vigor+Esteem Related Affect]. A lower score indicates overall better mood, while a lower score indicates worse overall mood

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Wilson, Ph.D., Principal Investigator — The Applied Science and Performance Institute
Locations (1):
- Applied Science and Performance Institute, Tampa, Florida, United States